CLINICAL TRIAL: NCT07146932
Title: Evaluating the Bambini Teens Exoskeleton for Pediatric Cerebral Palsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: COSMO ROBOTICS CO., Ltd (Industry)
Collaborators: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXO-CIP-002
Record Dates: First submitted 2025-08-13; First posted 2025-08-28 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy (CP)
Keywords: Bambini Teens; Cerebral Palsy; Exoskeleton; ExoAtlet; Cosmo Robotics; Wearable Robotic Devices
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Bambini Teens Exoskeleton Gait Training (Experimental): Participants in this arm will receive gait training using the Bambini Teens Exoskeleton. Each participant will complete six training sessions, each lasting 30 minutes, conducted 2-3 times per week over approximately 3 weeks.
  Interventions: Device: Pediatric Lower Limb Exoskeleton (Bambini Teens)

INTERVENTIONS:
Device: Pediatric Lower Limb Exoskeleton (Bambini Teens) — The Bambini Teens Exoskeleton is a wearable robotic device developed to assist lower limb movement and facilitate gait training for pediatric patients with mobility impairments such as cerebral palsy. The device provides powered assistance at the hip, knee, and ankle joints, supports adjustable gait parameters, and is designed for use in clinical rehabilitation settings under professional supervision.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and effectiveness of the Bambini Teens exoskeleton as a gait training tool in children aged 5 to 14 years diagnosed with cerebral palsy (CP). The main questions it aims to answer are:

* Is the Bambini Teens exoskeleton device safe and feasible as a gait training intervention for children with cerebral palsy, without resulting in a significant incidence of device-related serious adverse events?
* Is it feasible for physical therapists to use the Bambini Teens exoskeleton as a gait training intervention for children with cerebral palsy, meaning participants will successfully complete the training sessions?
* Will participants' mobility, specifically their self-selected walking speed, improve after receiving gait training using the Bambini Teens exoskeleton compared to baseline measurements?

Researchers will compare participants' mobility measured at baseline to their mobility after the intervention to see if improvements occur.

Participants will:

* Complete 6 gait training sessions using the Bambini Pediatric Exoskeleton, monitored by a licensed physical therapist.
* Each training session will be 30 minutes long, conducted 2-3 times per week for approximately 3 weeks.
* Undergo evaluations at baseline and post-intervention (after approximately 3 weeks), with each evaluation session lasting approximately 2 hours.
* May also participate in optional motor evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 5 and 14 years and diagnosed with cerebral palsy;
* have joint range of motion within normal functional limits for ambulation as determined by study staff;
* Be able and willing to comply with study procedures, including follow-up requirements;
* Patient cognitive status and ability to communicate must be at a level consistent with that required to participate in standard motor rehabilitation;
* can follow directions as determined by study staff;
* be able to physically fit into exoskeleton device; height from 110 to 160 cm (43 to 62 inches) and weighing up less than 65 kg (145 lbs);
* be able to walk 10 meters with the aid of a walking assistive device and/or a single human assistant;
* bilateral lower limb spasticity that allows lower limb range of motion within the device.

Exclusion Criteria:

* any medical issue that precludes full weight-bearing and ambulation (e.g. orthopedic injuries, pain, severe spasticity);
* skin issues that would prevent wearing the device;
* pre-existing condition that caused exercise intolerance;
* uncontrolled seizure disorder, spasticity or joint contracture that would interfere with walking;
* neuromuscular, neurological, cardiovascular or orthopedic pathologies that will interfere with neuromuscular function, ambulation, or limit the range of motion of the lower limbs;
* severe spasticity (Modified Ashworth Scale = or > 3);
* hip extension range of motion < 0 degrees, knee flexion contracture > 20 degrees, knee valgus > 40 degrees, 2 or more fractures within the past year, hip subluxation (> 40% migration),
* existing Baclofen pump, and/or Botox injections within the past 4 months of study enrollment;

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Device Safety | Baseline to end of intervention (approximately 3 weeks)
  Incidence of device-related serious adverse events (SAEs) and other adverse events (AEs) occurring during the intervention period, recorded in an adverse event log.
Participant Usage and Treatment Compliance | Baseline to end of intervention (approximately 3 weeks)
  Proportion of participants who complete all six planned gait training sessions under the supervision of a licensed physical therapist. Completion will be verified by session attendance and completion records.
Feasibility of Usage | Baseline to end of intervention (approximately 3 weeks)
  Proportion of participants for whom the treating physical therapist successfully fits the device and records session-specific device settings, as documented in the session logs.
Clinician Treatment Satisfaction | End of intervention (~3 weeks, at final assessment)
  Clinician satisfaction with the intervention, measured using a standardized FORM questionnaire completed by the treating physical therapist at the end of the intervention.

SECONDARY OUTCOMES:
Physical Impairment - Blood Pressure | Baseline to end of intervention (approximately 3 weeks)
  Change in resting systolic and diastolic blood pressure measured using a standard sphygmomanometer.
Physical Impairment - Muscle Strength | Baseline to end of intervention (approximately 3 weeks)
  Change in muscle strength of upper and lower limbs measured using the Manual Muscle Testing (MMT) scale (0-5 grades).
Physical Impairment - Joint Range of Motion | Baseline to end of intervention (approximately 3 weeks)
  Change in the range of motion of upper and lower limb joints measured using a goniometer, reported as change in degrees.
Physical Impairment - Spasticity | Baseline to end of intervention (approximately 3 weeks)
  Change in spasticity of lower extremities measured using the Modified Ashworth Scale (0-4 scores, with higher scores indicating greater spasticity).
Endurance | Baseline to end of intervention (approximately 3 weeks)
  Distance walked in meters during the 6-Minute Walk Test (6MWT), used as a submaximal test of aerobic capacity/endurance and a functional assessment of walking efficiency.
10-Meter Walk Test | Baseline to end of intervention (approximately 3 weeks)
  A functional ambulation assessment of walking speed over a 10-meter distance, reported in meters per second (m/s). Higher values indicate faster walking ability
Timed Up and Go (TUG) | Baseline to end of intervention (approximately 3 weeks)
  Assessment of functional mobility and balance, measuring the time (in seconds) required for a participant to stand up from a chair, walk 3 meters, turn, return, and sit down. Shorter times indicate better mobility.
Gait Mat Assessment | Baseline to end of intervention (approximately 3 weeks)
  Temporal and spatial gait parameters obtained from an instrumented walkway provide quantitative information about walking and standing balance. Values are reported in standard gait units (e.g., step length in cm, velocity in m/s).
Pediatric Balance Scale (PBS) | Baseline to end of intervention (approximately 3 weeks)
  A 14-item scale assessing functional balance in children, with scores ranging from 0 to 56. Higher scores indicate better balance.
Pediatric Quality of Life Inventory (PedsQL) | Baseline to end of intervention (approximately 3 weeks)
  Change in health-related quality of life assessed by the Pediatric Quality of Life Inventory (PedsQL). The PedsQL total score ranges from 0 to 100, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States